CLINICAL TRIAL: NCT02083653
Title: Open-label, Randomized, Controlled, Multicenter Phase II Trial Investigating 2 Sym004 Doses Versus Investigator's Choice (Best Supportive Care, Capecitabine, 5-FU) in Subjects With Metastatic Colorectal Cancer and Acquired Resistance to Anti-EGFR Monoclonal Antibodies
Brief Title: Sym004 vs Standard of Care in Subjects With Metastatic Colorectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Symphogen A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Sym004-05; 2013-003829-29 (EudraCT Number); EMR200637-002 (Other: Merck KGaA)
Record Dates: First submitted 2014-03-07; First posted 2014-03-11 (Estimated); Results first posted 2018-12-24 (Actual); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Metastatic Colorectal Cancer
Keywords: Metastatic Colorectal Cancer; Best Supportive Care; Capecitabine; Fluorouracil (5-FU); Sym004
MeSH Terms: conditions — Colorectal Neoplasms | interventions — futuximab; Fluorouracil; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm A: Sym004 (12 mg/kg) (Experimental): Sym004 will be administered as an intravenous infusion at a dose of 12 milligrams per kilogram (mg/kg) weekly until unacceptable toxicity, disease progression, or consent withdrawal.
  Interventions: Drug: Sym004 (12 mg/kg)
- Arm B: Sym004 (9/6 mg/kg) (Experimental): Sym004 will be administered as an intravenous infusion at a loading dose of 9 mg/kg followed by 6 mg/kg weekly until unacceptable toxicity, disease progression, or consent withdrawal.
  Interventions: Drug: Sym004 (9/6 mg/kg)
- Arm C: Investigator's Choice (Active Comparator): Best supportive care (BSC) or Fluorouracil (5-FU) or Capecitabine will be given as per Investigator's discretion.
  Interventions: Other: Best Supportive Care (BSC); Drug: Fluorouracil (5-FU); Drug: Capecitabine

INTERVENTIONS:
Drug: Sym004 (12 mg/kg) — Sym004 is a 1:1 mixture of two mAbs (futuximab and modotuximab) which bind to two non-overlapping epitopes of the EGFR.
  Arms: Arm A: Sym004 (12 mg/kg)
Drug: Sym004 (9/6 mg/kg) — Sym004 is a 1:1 mixture of two mAbs (futuximab and modotuximab) which bind to two non-overlapping epitopes of the EGFR.
  Arms: Arm B: Sym004 (9/6 mg/kg)
Other: Best Supportive Care (BSC) — BSC is the best palliative care as per Investigator's discretion, excluding antineoplastic agents. BSC may include, but is not limited to, antibiotics, analgesics, antiemetics, blood transfusions, and nutritional support.
  Arms: Arm C: Investigator's Choice
Drug: Fluorouracil (5-FU) — 5-FU will be administered at doses and schedules as per Investigator's discretion and in line with the local package insert.
  Other Names: Adrucil
  Arms: Arm C: Investigator's Choice
Drug: Capecitabine — Capecitabine will be administered at doses and schedules as per Investigator's discretion and in line with the local package insert.
  Other Names: Xeloda
  Arms: Arm C: Investigator's Choice

SUMMARY:
This is a Phase 2, open-label, randomized, 3-arm trial investigating the efficacy of two Sym004 doses (Arm A and Arm B) compared with a control group (Arm C) in subjects with metastatic colorectal cancer (mCRC) and acquired resistance to anti-epidermal growth factor receptor (EGFR) monoclonal antibodies (mAbs).

DETAILED DESCRIPTION:
This trial assesses the efficacy of two different weekly dosing regimens of Sym004 (Arm A: 12 mg/kg/week versus Arm B: 9 mg/kg loading dose followed by 6 mg/kg/week) compared with investigator's choice in terms of overall survival time in subjects with mCRC. Subjects assigned to Arm C will receive best supportive care (BSC), Fluorouracil (5-FU), or Capecitabine, per local standard of care.

Subjects will receive treatment until unacceptable toxicity, disease progression, withdrawal of consent, or until the subject meets any of the criteria for treatment discontinuation or trial discontinuation. Therefore, the duration of treatment will differ among individuals and cannot be fixed in advance.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent obtained before undergoing any study-related activities
* Male or female, at least 18 years of age
* Subjects with histologically or cytologically confirmed mCRC, Kirsten rat sarcoma wild-type (KRAS WT) at initial diagnosis
* Failure of or intolerance to 5-FU, Oxaliplatin, and Irinotecan
* Acquired resistance to marketed anti-EGFR mAbs as defined in the protocol
* Measurable disease defined as one or more target lesions according to RECIST
* Life expectancy of at least 3 months
* Eastern Cooperative Oncology Group (ECOG) performance status less than or equal to 1
* Other protocol defined inclusion criteria could apply

Exclusion Criteria:

* Pretreatment with regorafenib.
* Subjects who in the opinion of the subject and investigator would benefit more from regorafenib treatment (except where regorafenib is not reimbursed in the country)
* Skin rash Common Terminology Criteria for AEs (CTCAE) Grade greater than 1 from previous anti-EGFR therapy at time of randomization
* Magnesium less than 0.9 milligram per deciliter (mg/dL)
* Known hypersensitivity to any of the treatment ingredients. Known previous Grade 3-4 infusion related reactions with anti-EGFR mABs
* Other protocol defined exclusion criteria could apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 254 (Actual)
Dates: Start 2014-03-06 (Actual); Primary Completion 2016-10-24 (Actual); Study Completion 2017-04-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Josep Tabernero, MD, PhD, Principal Investigator — Vall d'Hebron University Hospital
Locations (54):
- United States (9):
  - USC Norris Comprehensive Cancer Center, Los Angeles, California
  - Sharp Memorial Hospital, San Diego, California
  - Florida Cancer Specialists-Broadway, Fort Myers, Florida
  - Hematology - Oncology Associates of Treasure Coast, Port Saint Lucie, Florida
  - Florida Cancer Specialists, St. Petersburg, Florida
  - Mercy Research, Springfield, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Comprehensive Cancer Centers of Nevada, Henderson, Nevada
  - Texas Oncology, P.A., Tyler, Texas
- SMZ Süd - Kaiser Franz Josef Spital Wien, Vienna, Austria
- Belgium (7):
  - ULB Hôpital Erasme, Brussels
  - Cliniques Universitaires Saint-Luc, Brussels
  - Universitair Ziekenhuis Gent, Ghent
  - UZ Leuven, Leuven
  - CHU Ambroise Paré, Mons
  - Clinique et Maternité Sainte-Elisabeth, Namur
  - CHU Mont-Godinne, Yvoir
- France (8):
  - ICO - Site Paul Papin, Angers
  - Institut Sainte Catherine, Avignon
  - Groupe Hospitalier Saint André - Hôpital Saint André, Bordeaux
  - Centre Georges François Leclerc, Dijon
  - Centre Léon Bérard, Lyon
  - CRLCC Eugene Marquis, Rennes
  - ICO - Site René Gauducheau, Saint-Herblain
  - CHU de Toulouse - Hôpital Rangueil, Toulouse
- Germany (2):
  - Universitaetsklinikum Carl Gustav Carus TU Dresden, Dresden
  - Klinikum der Johann Wolfgang Goethe-Universitaet, Frankfurt
- Hungary (4):
  - Uzsoki Utcai Korhaz, Budapest
  - Borsod-Abauj-Zemplen Megyei Korhaz es Egyetemi Oktato Korhaz, Miskolc
  - SzSzB Megyei Korhazak es Egyetemi Oktatokorhaz, Nyíregyháza
  - Jasz-Nagykun-Szolnok Megyei Korhaz-Rendelointezet, Szolnok
- Italy (9):
  - Azienda Ospedaliero Universitaria Ospedali Riuniti, Ancona
  - Azienda Ospedaliero Universitaria San Martino, Genova
  - Azienda Ospedaliera Ospedale Niguarda Ca' Granda, Milan
  - Seconda Università degli Studi di Napoli, Napoli
  - IOV - Istituto Oncologico Veneto IRCCS, Padua
  - Azienda Ospedaliero Universitaria Pisana, Pisa
  - Policlinico Universitario Agostino Gemelli, Roma
  - Presidio Ospedaliero SS. Trinità Sora, Sora
  - Azienda Ospedaliera S. Maria Di Terni, Terni
- Poland (4):
  - SPZOZ MSW zWarmińsko-MazurskimCen.Onko.wOlsztynie, Olsztyn
  - Wielkopolskie Centrum Onkologii, Poznan
  - Wojewodzki Szpital Zespolony im. L. Rydygiera w Toruniu, Torun
  - Centrum Onkologii-Instytut im. M. Sklodowskiej Curie, Warsaw
- Russia (2):
  - BHI of Omsk region "Clinical Oncology Dispensary", Omsk
  - St. Petersburg SHI "City Clinical Oncology Dispensary", Saint Petersburg
- Spain (8):
  - Hospital del Mar, Barcelona
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Clinic i Provincial de Barcelona, Barcelona
  - ICO l´Hospitalet - Hospital Duran i Reynals, Barcelona
  - Hospital General Universitario Gregorio Marañon, Madrid
  - Centro Integral Oncologico Clara Campal, Madrid
  - Hospital Universitario Central de Asturias, Oviedo
  - Hospital Universitario Virgen del Rocio, Seville

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Aaronson NK, Ahmedzai S, Bergman B, Bullinger M, Cull A, Duez NJ, Filiberti A, Flechtner H, Fleishman SB, de Haes JC, et al. The European Organization for Research and Treatment of Cancer QLQ-C30: a quality-of-life instrument for use in international clinical trials in oncology. J Natl Cancer Inst. 1993 Mar 3;85(5):365-76. doi: 10.1093/jnci/85.5.365. PMID 8433390
- [Background] Fayers PM, Aaronson NK, Bjordal K, Groenvold M, Curran D, Bottomley A, on behalf of the EORTC Quality of Life Group. The EORTC QLQ-C30 Scoring Manual (3rd Edition). Published by: European Organisation for Research and Treatment of Cancer, Brussels 2001.

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm A: Sym004 (12 mg/kg): Sym004 will be administered as an intravenous infusion at a dose of 12 milligrams per kilogram (mg/kg) weekly until unacceptable toxicity, disease progression, or consent withdrawal.
  Sym004 (12 mg/kg): Sym004 is a 1:1 mixture of two monoclonal antibodies (mAbs) (futuximab and modotuximab) which bind to two non-overlapping epitopes of the epidermal growth factor receptor (EGFR).
Period: Overall Study
Arm/Group | Arm A: Sym004 (12 mg/kg) | Arm B: Sym004 (9/6 mg/kg) | Arm C: Investigator's Choice
Started | 83 | 86 | 85
Completed | 1 | 1 | 1
Not Completed | 82 | 85 | 84
Not completed — Randomized but not Treated | 0 | 2 | 7
Not completed — Adverse Event | 12 | 5 | 4
Not completed — Lost to Follow-up | 1 | 0 | 0
Not completed — Death | 2 | 2 | 2
Not completed — Progressive Disease | 65 | 73 | 63
Not completed — Withdrawal by Subject | 2 | 1 | 2
Not completed — Other Events | 0 | 2 | 2
Not completed — Reason Missing | 0 | 0 | 4

BASELINE CHARACTERISTICS:
Population: The baseline analysis population was the intent-to-treat (ITT) analysis set.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A: Sym004 (12 mg/kg) | Arm B: Sym004 (9/6 mg/kg) | Arm C: Investigator's Choice | Total
Number analyzed (Participants) | 83 | 86 | 85 | 254
Age, Continuous [Mean (Standard Deviation); unit: years] — Age is relative to time of informed consent for this trial. Population: The age summary does not include subjects living in Germany.
  years
    number analyzed (Participants) | 79 | 86 | 84 | 249
    (all) | 62.2 (9.91) | 64.2 (10.41) | 61.4 (10.70) | 62.6 (10.38)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 32 | 31 | 94
  Male | 52 | 54 | 54 | 160
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Ethnicity is presented as 'Not Reported' for subjects living in France.
  Participants
    Hispanic or Latino | 5 | 5 | 5 | 15
    Not Hispanic or Latino | 69 | 72 | 70 | 211
    Unknown or Not Reported | 9 | 9 | 10 | 28
Race (NIH/OMB) [Count of Participants; unit: Participants] — Race is presented as 'Not Reported' for subjects living in France.
  Participants
    American Indian or Alaska Native | 0 | 0 | 0 | 0
    Asian | 1 | 0 | 0 | 1
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
    Black or African American | 1 | 2 | 0 | 3
    White | 72 | 75 | 73 | 220
    More than one race | 0 | 0 | 0 | 0
    Unknown or Not Reported | 9 | 9 | 12 | 30
Region of Enrollment [Number; unit: participants]
  Austria | 0 | 1 | 1 | 2
  Belgium | 3 | 6 | 5 | 14
  Hungary | 0 | 1 | 5 | 6
  United States | 8 | 6 | 8 | 22
  Poland | 10 | 8 | 7 | 25
  Italy | 17 | 12 | 20 | 49
  France | 9 | 9 | 10 | 28
  Germany | 4 | 0 | 1 | 5
  Russia | 8 | 12 | 10 | 30
  Spain | 24 | 31 | 18 | 73
Height [Mean (Standard Deviation); unit: centimeters (cm)] | 168.9 (10.82) | 169.1 (9.71) | 167.9 (9.56) | 168.7 (10.01)
Weight [Mean (Standard Deviation); unit: kilograms (kg)] | 75.3 (13.51) | 74.0 (14.14) | 76.0 (16.13) | 75.1 (14.61)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 26.5 (4.43) | 25.8 (4.26) | 26.8 (4.59) | 26.4 (4.43)

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS) Time
Description: OS based on product-limit (Kaplan-Meier) estimates. Confidence intervals for the median are calculated according to Brookmeyer and Crowley.
  If a subject had not died, survival time was censored at the last date the subject was known to be alive.
Time Frame: From randomization until the date of death (assessed up to 32 months).
Population: The analysis population was the intent-to-treat (ITT) subpopulation, which includes all subjects who were randomized to investigational medicinal product (IMP). Analyses performed on the ITT analysis set will take into account subjects' allocation to treatment groups as randomized and not as treated.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A: Sym004 (12 mg/kg) | Arm B: Sym004 (9/6 mg/kg) | Arm C: Investigator's Choice
Number analyzed (Participants) | 83 | 86 | 85
months | 7.9 [6.5 to 9.9] | 10.3 [9.0 to 12.9] | 9.6 [8.3 to 12.2]

2. Secondary Outcome: Best Overall Response (OR) According to the Response Evaluation Criteria In Solid Tumors Version 1.1 (RECIST v1.1)
Description: Tumor assessments were done via computed tomography (CT) or magnetic resonance imaging (MRI) scans and evaluated per RECIST v1.1. The assessment for measurable disease during screening (within 14 days prior to Day 1) acts as the baseline assessment. Best OR was summarized for each treatment group by means of counts and percentages for the following categories: Complete Response (CR: disappearance of all target lesions), Partial Response (PR: at least a 30% decrease in the sum of diameters of target lesions), Progressive Disease (PD: at least a 20% increase in the sum of diameters of target lesions), Stable Disease (SD: neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD) or Not Evaluable (NE).
Time Frame: From randomization until first radiological confirmed or clinical progression event, or death due to any cause, within 12 weeks after last tumor assessment (assessed up to 32 months).
Population: The analysis population was the ITT subpopulation, which includes all subjects who were randomized to IMP. Analyses performed on the ITT analysis set will take into account subjects' allocation to treatment groups as randomized and not as treated.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: Sym004 (12 mg/kg) | Arm B: Sym004 (9/6 mg/kg) | Arm C: Investigator's Choice
Number analyzed (Participants) | 83 | 86 | 85
Participants
  Complete Response (CR) | 0 | 0 | 1
  Partial Response (PR) | 11 | 8 | 1
  Stable Disease (SD) | 40 | 47 | 37
  Progressive Disease (PD) | 27 | 28 | 31
  Not Evaluable (NE) | 5 | 3 | 15

3. Secondary Outcome: Progression Free Survival (PFS) Time
Description: PFS based on product-limit (Kaplan-Meier) estimates. Confidence intervals for the median are calculated according to Brookmeyer and Crowley. Death will only be considered as an event if it occurs within 12 weeks after last tumor response assessment without progression.
Time Frame: From randomization until first event, where an event can be a progression (radiological confirmed or clinical progression) or death due to any cause (assessed up to 32 months).
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A: Sym004 (12 mg/kg) | Arm B: Sym004 (9/6 mg/kg) | Arm C: Investigator's Choice
Number analyzed (Participants) | 83 | 86 | 85
months | 2.8 [1.8 to 3.2] | 2.7 [2.6 to 3.3] | 2.6 [1.4 to 3.1]

4. Secondary Outcome: Time to Treatment Failure (TTF)
Description: TTF based on product-limit (Kaplan-Meier) estimates. Confidence intervals for the median are calculated according to Brookmeyer and Crowley.
Time Frame: From randomization until treatment discontinuation for any reason, including disease progression or death (assessed up to 32 months).
Population: The analysis population was the ITT subpopulation, which includes all subjects who were randomized to IMP. Analyses performed on the ITT analysis set will take into account subjects' allocation to treatment groups as randomized and not as treated. Subjects who were randomized but not treated have been censored at the date of randomization.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A: Sym004 (12 mg/kg) | Arm B: Sym004 (9/6 mg/kg) | Arm C: Investigator's Choice
Number analyzed (Participants) | 83 | 86 | 85
months | 2.1 [1.4 to 2.7] | 2.6 [2.2 to 2.6] | 1.6 [1.2 to 2.7]

5. Secondary Outcome: Occurrence and Nature of Adverse Events (AEs), as Assessed by the Common Terminology Criteria for AEs (Version 4.03) (CTCAE v4.03).
Description: AEs were coded according to the Medical Dictionary for Regulatory Activities (MedDRA) classification. The incidence and type of AEs (i.e., serious AE [SAE], treatment-emergent AE [TEAE]) were summarized by dose cohort according to MedDRA system organ classes and preferred terms. An AE was considered as treatment-emergent if it occurred during or after the first IMP administration. An AE that occurred before the first IMP administration and worsened thereafter was also considered an AE. Worsening was reported as a new AE.
Time Frame: From Baseline up to 28 days after the last IMP administration.
Population: The analysis population was the safety analysis subpopulation, which includes all subjects who were administered any dose of IMP, and in addition those subjects in Arm C for which the intended control treatment is BSC. Subjects will be analyzed as treated and not as randomized.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: Sym004 (12 mg/kg) | Arm B: Sym004 (9/6 mg/kg) | Arm C: Investigator's Choice
Number analyzed (Participants) | 83 | 84 | 78
Participants
  At least one TEAE | 83 | 84 | 67
  At least one Serious TEAE | 27 | 23 | 12
  TEAE leading to dose reduction | 29 | 17 | 8
  TEAE leading to interruption of trial treatment | 58 | 47 | 10
  TEAE leading to trial treatment withdrawal | 12 | 5 | 6
  TEAE related to trial treatment | 81 | 80 | 46
  TEAE, Grade >=3 | 67 | 53 | 25
  Dermatologic toxicity | 78 | 78 | 8
  Infusion-related reaction | 27 | 26 | 0
  TEAE resulting in death | 4 | 4 | 3
  Related Serious TEAE | 9 | 6 | 2
  Related TEAE leading to dose reduction | 29 | 17 | 6
  Related TEAE leading to interruption of treatment | 53 | 42 | 7
  Related TEAE leading to treatment withdrawal | 9 | 2 | 3
  Related TEAE, Grade >=3 | 58 | 41 | 9
  Related TEAE resulting in death | 0 | 0 | 0

6. Secondary Outcome: Relative Dose Intensity of Sym004
Description: Treatment duration (weeks) is calculated as [(last dose date of Sym004 - first dose date of Sym004)+7] / 7 days.
  Sym004 dose received (mg/kg) is calculated as (total dose administered (mg)/weight (kg)).
  Dose Intensity is calculated as (cumulative Sym004 dose (mg/kg) / treatment duration (weeks)).
  Relative Dose Intensity is calculated as (dose intensity / planned dose intensity at randomization)*100.
  Percentages are based on the number of subjects in the safety analysis set.
Time Frame: From first dose of study drug until disease progression (assessed up to 32 months).
Population: The analysis population was the safety analysis subpopulation, which includes all subjects who were administered any dose of IMP. Subjects will be analyzed as treated and not as randomized.
Measure: Mean (Standard Deviation); unit: percentage of relative dose intensity
Arm/Group | Arm A: Sym004 (12 mg/kg) | Arm B: Sym004 (9/6 mg/kg)
Number analyzed (Participants) | 83 | 84
percentage of relative dose intensity | 80.49 (20.020) | 88.91 (13.843)

7. Secondary Outcome: Pharmacokinetic (PK) Parameters: Sym004 Concentrations
Description: The Sym004 serum concentration used for the PK evaluation was calculated as the sum of the serum concentrations of the 2 component monoclonal antibodies of Sym004 (futuximab and modotuximab).
  Trough Concentration (Ctrough) is equivalent to the concentration collected at the pre-dose timepoint.
  Maximum Concentration (Cmax) is equivalent to the concentration collected at the end of infusion (EOI) timepoint.
Time Frame: Weeks 3, 5, and 7 and at the End of Treatment visit, including a Week 1 and Week 2 subset.
Population: The analysis population was the PK analysis set. Bioanalysis for serum concentration was done for a subset of subjects (N=19) at all scheduled timepoints; it was carried out only at Weeks 3, 5, 7 and the End of Treatment visit for all other subjects. Additionally, the Week 1 Day 1 EOI concentration for Subject 2740012 was assessed.
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | Arm A: Sym004 (12 mg/kg) | Arm B: Sym004 (9/6 mg/kg)
Number analyzed (Participants) | 80 | 83
ug/mL
  Screening (Pre-dose): number analyzed (Participants) | 11 | 8
  Screening (Pre-dose) | 0.50 (0.000) | 0.50 (0.000)
  Week 1 Day 1 (Pre-dose): number analyzed (Participants) | 11 | 8
  Week 1 Day 1 (Pre-dose) | 0.50 (0.000) | 0.75 (0.700)
  Week 1 Day 1 (EOI): number analyzed (Participants) | 12 | 8
  Week 1 Day 1 (EOI) | 182.95 (97.686) | 174.44 (47.023)
  Week 1 Day 1 (0.5 hours after EOI): number analyzed (Participants) | 11 | 8
  Week 1 Day 1 (0.5 hours after EOI) | 214.98 (46.242) | 184.84 (33.103)
  Week 1 Day 1 (1 hour after EOI): number analyzed (Participants) | 11 | 8
  Week 1 Day 1 (1 hour after EOI) | 209.80 (60.707) | 189.24 (38.923)
  Week 1 Day 1 (2 hours after EOI): number analyzed (Participants) | 11 | 8
  Week 1 Day 1 (2 hours after EOI) | 197.31 (65.801) | 181.68 (37.577)
  Week 1 Day 1 (4 hours after EOI): number analyzed (Participants) | 11 | 8
  Week 1 Day 1 (4 hours after EOI) | 188.75 (68.421) | 171.63 (35.862)
  Week 2 Day 1 (Pre-dose): number analyzed (Participants) | 11 | 8
  Week 2 Day 1 (Pre-dose) | 45.37 (28.604) | 38.76 (10.311)
  Week 2 Day 1 (EOI): number analyzed (Participants) | 11 | 8
  Week 2 Day 1 (EOI) | 275.42 (80.975) | 145.91 (47.950)
  Week 3 Day 1 (Pre-dose): number analyzed (Participants) | 76 | 80
  Week 3 Day 1 (Pre-dose) | 92.66 (38.443) | 44.26 (20.995)
  Week 3 Day 1 (EOI): number analyzed (Participants) | 73 | 79
  Week 3 Day 1 (EOI) | 323.35 (83.412) | 170.18 (50.323)
  Week 5 Day 1 (Pre-dose): number analyzed (Participants) | 58 | 63
  Week 5 Day 1 (Pre-dose) | 125.73 (61.644) | 49.26 (30.252)
  Week 5 Day 1 (EOI): number analyzed (Participants) | 56 | 63
  Week 5 Day 1 (EOI) | 354.91 (108.263) | 168.94 (67.901)
  Week 7 Day 1 (Pre-dose): number analyzed (Participants) | 41 | 55
  Week 7 Day 1 (Pre-dose) | 128.30 (77.437) | 58.38 (47.505)
  Week 7 Day 1 (EOI): number analyzed (Participants) | 37 | 53
  Week 7 Day 1 (EOI) | 346.83 (136.083) | 163.11 (74.967)
  End of Treatment: number analyzed (Participants) | 57 | 55
  End of Treatment | 64.55 (79.250) | 17.61 (24.474)

8. Secondary Outcome: Pharmacokinetic (PK) Parameters: Time of Maximum Plasma Concentration (Tmax)
Description: Tmax was defined as the time the PK sample was taken at end of infusion (EOI) relative to the start time of infusion (i.e., time between the start of infusion and the time of the EOI sample). For presentation of individual PK parameters and calculation of mean parameters, half of the lower limit of quantitation (LLOQ) value was used for concentration values below the LLOQ. The Sym004 serum concentration used for the PK evaluation was calculated as the sum of the serum concentrations of the 2 component monoclonal antibodies of Sym004, futuximab and modotuximab.
Time Frame: Day 1 on Weeks 1-3 followed by Week 5 Day 1 and Week 7 Day 1.
Population: The analysis population was the PK analysis set, defined as subjects having at least 1 Sym004 serum concentration above the LLOQ. Exposure to Sym004 was confirmed in the majority of subjects treated with Sym004 for at least 1 timepoint post-dose.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Arm A: Sym004 (12 mg/kg) | Arm B: Sym004 (9/6 mg/kg)
Number analyzed (Participants) | 80 | 83
hours
  Week 1 Day 1: number analyzed (Participants) | 12 | 8
  Week 1 Day 1 | 3.14 (0.822) | 2.79 (0.210)
  Week 2 Day 1: number analyzed (Participants) | 11 | 8
  Week 2 Day 1 | 2.82 (0.306) | 2.33 (0.459)
  Week 3 Day 1: number analyzed (Participants) | 72 | 79
  Week 3 Day 1 | 3.01 (0.555) | 2.34 (0.477)
  Week 5 Day 1: number analyzed (Participants) | 56 | 63
  Week 5 Day 1 | 2.74 (0.532) | 2.06 (0.448)
  Week 7 Day 1: number analyzed (Participants) | 37 | 52
  Week 7 Day 1 | 2.83 (0.867) | 2.06 (0.473)

9. Secondary Outcome: Host Immune Response: Number of Subjects With Anti-drug Antibodies (ADAs) to Sym004 Over Time
Description: A validated double antigen bridging ELISA was used for screening, confirmation, and titration of patient samples for anti-Sym004 ADA. Using rabbit anti-Sym004 as an ADA control antibody, the lower limit of detection was 54 ng/mL in the absence of Sym004 and 500 ng/mL in the presence of Sym004 at 5 µg/mL The timepoints for ADA sampling were chosen by the original sponsor for this trial. After the trial was transferred to Symphogen A/S, it was determined that not all samples were necessary for analysis. This is why the collection time points specified in the Outcome Measure Time Frame do not match with the Outcome Measure Data Table.
Time Frame: Every two weeks (Days 15, 29, and 43) followed by every six weeks thereafter (Days 78, 120, 162, etc.) until the End of Treatment Visit
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: Sym004 (12 mg/kg) | Arm B: Sym004 (9/6 mg/kg)
Number analyzed (Participants) | 83 | 84
Participants
  Screening: Negative | 78 | 81
  Screening: Positive | 2 | 0
  Screening: Not Reportable | 1 | 0
  Screening: Missing | 2 | 3
  Week 5 Day 1: Negative | 59 | 62
  Week 5 Day 1: Positive | 0 | 0
  Week 5 Day 1: Not Reportable | 0 | 0
  Week 5 Day 1: Missing | 24 | 22
  Week 12: Negative | 24 | 35
  Week 12: Positive | 0 | 0
  Week 12: Not Reportable | 0 | 0
  Week 12: Missing | 59 | 49
  Week 13: Negative | 1 | 1
  Week 13: Positive | 0 | 0
  Week 13: Not Reportable | 0 | 0
  Week 13: Missing | 82 | 83
  Week 24: Negative | 0 | 1
  Week 24: Positive | 0 | 0
  Week 24: Not Reportable | 0 | 0
  Week 24: Missing | 83 | 83
  End of Treatment Visit: Negative | 60 | 55
  End of Treatment Visit: Positive | 0 | 0
  End of Treatment Visit: Not Reportable | 0 | 0
  End of Treatment Visit: Missing | 23 | 29

10. Secondary Outcome: Quality of Life Assessed by the EORTC QLQ-C30 (Version 3)
Description: Scale: European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (Version 3) [QLQ-C30, Version 3].
  The QLQ-C30 is a 30-question scale used to assess cancer patients' quality of life based on 15 factors (e.g., global health status, physical functioning, role functioning, etc.). The scale is composed of both multi-item scales and single-item measures. All of the scales and single-item measures range in score from 0 to 100:
  * A high score for a functional scale represents a healthy level of functioning.
  * A high score for the global health status represents a high quality of life.
  * A high score for a symptom scale/item represents a high level of symptomatology (problems).
Time Frame: Assessed every 6 weeks (week 1 and week 7 reported)
Population: This measure was self-reported. Numbers analyzed between Week 1 and Week 7 differ from each other, as well from the overall number of subjects analyzed. Data could not be collected from subjects not compliant with reporting or once discontinued.
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Arm A: Sym004 (12 mg/kg) | Arm B: Sym004 (9/6 mg/kg) | Arm C: Investigator's Choice
Number analyzed (Participants) | 83 | 86 | 85
score on a scale
  Global Health Status (Week 1 Day 1): number analyzed (Participants) | 74 | 79 | 66
  Global Health Status (Week 1 Day 1) | 55.5 [0 to 92] | 59.7 [8 to 100] | 55.8 [8 to 100]
  Global Health Status (Week 7 Day 1): number analyzed (Participants) | 48 | 48 | 36
  Global Health Status (Week 7 Day 1) | 57.4 [25 to 100] | 59.4 [17 to 100] | 59.7 [17 to 100]
  Physical Functioning (Week 1 Day 1): number analyzed (Participants) | 75 | 81 | 69
  Physical Functioning (Week 1 Day 1) | 76.4 [7 to 100] | 78.7 [27 to 100] | 77.7 [27 to 100]
  Physical Functioning (Week 7 Day 1): number analyzed (Participants) | 51 | 49 | 36
  Physical Functioning (Week 7 Day 1) | 82.1 [13 to 100] | 83.0 [47 to 100] | 76.7 [40 to 100]
  Role Functioning (Week 1 Day 1): number analyzed (Participants) | 76 | 81 | 69
  Role Functioning (Week 1 Day 1) | 75.0 [0 to 100] | 76.4 [0 to 100] | 72.5 [0 to 100]
  Role Functioning (Week 7 Day 1): number analyzed (Participants) | 51 | 49 | 36
  Role Functioning (Week 7 Day 1) | 81.1 [33 to 100] | 82.4 [50 to 100] | 72.8 [17 to 100]
  Emotional Functioning (Week 1 Day 1): number analyzed (Participants) | 73 | 79 | 67
  Emotional Functioning (Week 1 Day 1) | 76.6 [17 to 100] | 77.8 [17 to 100] | 73.2 [0 to 100]
  Emotional Functioning (Week 7 Day 1): number analyzed (Participants) | 49 | 48 | 36
  Emotional Functioning (Week 7 Day 1) | 74.8 [0 to 100] | 82.7 [33 to 100] | 75.3 [17 to 100]
  Cognitive Functioning (Week 1 Day 1): number analyzed (Participants) | 74 | 79 | 67
  Cognitive Functioning (Week 1 Day 1) | 87.4 [33 to 100] | 86.2 [17 to 100] | 87.5 [50 to 100]
  Cognitive Functioning (Week 7 Day 1): number analyzed (Participants) | 49 | 48 | 36
  Cognitive Functioning (Week 7 Day 1) | 88.1 [33 to 100] | 88.5 [33 to 100] | 87.0 [33 to 100]
  Social Functioning (Week 1 Day 1): number analyzed (Participants) | 74 | 79 | 67
  Social Functioning (Week 1 Day 1) | 78.2 [17 to 100] | 80.2 [17 to 100] | 75.4 [17 to 100]
  Social Functioning (Week 7 Day 1): number analyzed (Participants) | 49 | 48 | 36
  Social Functioning (Week 7 Day 1) | 77.9 [0 to 100] | 83.4 [50 to 100] | 72.7 [0 to 100]
  Fatigue Symptoms (Week 1 Day 1): number analyzed (Participants) | 75 | 81 | 69
  Fatigue Symptoms (Week 1 Day 1) | 35.3 [0 to 89] | 32.2 [0 to 100] | 34.7 [0 to 100]
  Fatigue Symptoms (Week 7 Day 1): number analyzed (Participants) | 51 | 49 | 36
  Fatigue Symptoms (Week 7 Day 1) | 26.3 [0 to 78] | 25.3 [0 to 78] | 33.2 [0 to 78]
  Nausea & Vomiting Symptoms (Week 1 Day 1): number analyzed (Participants) | 76 | 81 | 69
  Nausea & Vomiting Symptoms (Week 1 Day 1) | 7.9 [0 to 67] | 6.4 [0 to 100] | 7.8 [0 to 83]
  Nausea & Vomiting Symptoms (Week 7 Day 1): number analyzed (Participants) | 51 | 49 | 36
  Nausea & Vomiting Symptoms (Week 7 Day 1) | 5.6 [0 to 33] | 5.1 [0 to 50] | 8.4 [0 to 50]
  Pain Symptoms (Week 1 Day 1): number analyzed (Participants) | 76 | 81 | 69
  Pain Symptoms (Week 1 Day 1) | 27.2 [0 to 100] | 23.6 [0 to 100] | 27.8 [0 to 100]
  Pain Symptoms (Week 7 Day 1): number analyzed (Participants) | 50 | 49 | 36
  Pain Symptoms (Week 7 Day 1) | 12.7 [0 to 50] | 14.6 [0 to 67] | 24.1 [0 to 83]
  Dyspnoea Symptoms (Week 1 Day 1): number analyzed (Participants) | 75 | 81 | 69
  Dyspnoea Symptoms (Week 1 Day 1) | 15.9 [0 to 100] | 17.2 [0 to 100] | 16.4 [0 to 100]
  Dyspnoea Symptoms (Week 7 Day 1): number analyzed (Participants) | 51 | 49 | 36
  Dyspnoea Symptoms (Week 7 Day 1) | 10.4 [0 to 67] | 8.8 [0 to 100] | 15.7 [0 to 100]
  Insomnia Symptoms (Week 1 Day 1): number analyzed (Participants) | 76 | 80 | 69
  Insomnia Symptoms (Week 1 Day 1) | 29.3 [0 to 100] | 19.1 [0 to 100] | 21.7 [0 to 100]
  Insomnia Symptoms (Week 7 Day 1): number analyzed (Participants) | 51 | 49 | 36
  Insomnia Symptoms (Week 7 Day 1) | 27.4 [0 to 100] | 16.9 [0 to 100] | 16.6 [0 to 67]
  Appetite Loss Symptoms (Week 1 Day 1): number analyzed (Participants) | 76 | 81 | 69
  Appetite Loss Symptoms (Week 1 Day 1) | 22.3 [0 to 100] | 17.6 [0 to 100] | 22.2 [0 to 100]
  Appetite Loss Symptoms (Week 7 Day 1): number analyzed (Participants) | 51 | 49 | 36
  Appetite Loss Symptoms (Week 7 Day 1) | 16.9 [0 to 100] | 17.5 [0 to 67] | 23.0 [0 to 100]
  Constipation Symptoms (Week 1 Day 1): number analyzed (Participants) | 73 | 79 | 67
  Constipation Symptoms (Week 1 Day 1) | 15.0 [0 to 67] | 16.0 [0 to 100] | 11.4 [0 to 100]
  Constipation Symptoms (Week 7 Day 1): number analyzed (Participants) | 49 | 48 | 36
  Constipation Symptoms (Week 7 Day 1) | 11.5 [0 to 67] | 8.3 [0 to 67] | 11.1 [0 to 67]
  Diarrhoea Symptoms (Week 1 Day 1): number analyzed (Participants) | 74 | 78 | 67
  Diarrhoea Symptoms (Week 1 Day 1) | 12.5 [0 to 100] | 8.5 [0 to 100] | 15.9 [0 to 100]
  Diarrhoea Symptoms (Week 7 Day 1): number analyzed (Participants) | 49 | 48 | 36
  Diarrhoea Symptoms (Week 7 Day 1) | 8.8 [0 to 100] | 11.1 [0 to 67] | 11.0 [0 to 67]
  Financial Difficulties (Week 1 Day 1): number analyzed (Participants) | 74 | 78 | 67
  Financial Difficulties (Week 1 Day 1) | 19.7 [0 to 67] | 16.6 [0 to 100] | 23.3 [0 to 100]
  Financial Difficulties (Week 7 Day 1): number analyzed (Participants) | 48 | 48 | 36
  Financial Difficulties (Week 7 Day 1) | 19.4 [0 to 100] | 15.2 [0 to 67] | 19.3 [0 to 100]

11. Secondary Outcome: Quality of Life Assessed by EORTC QLQ-CR29
Description: Scale: European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire - Colorectal Cancer Module (QLQ-CR29).
  The QLQ-CR29 is a 29-question scale used to assess colorectal cancer patients' quality of life based on 22 factors (e.g., body image, anxiety, weight, etc.). The scale is composed of both multi-item scales and single-item measures. All of the scales and single-item measures range in score from 0 to 100:
  * A high score for a functional scale/item represents an unhealthy level of functioning, with the exception of one (1) scale pertaining to sexual interest (separated by sex).
  * A high score for a symptom scale/item represents a high level of symptomatology (problems).
Time Frame: Assessed every 6 weeks (week 1 and week 7 reported)
Population: as for outcome 10
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Arm A: Sym004 (12 mg/kg) | Arm B: Sym004 (9/6 mg/kg) | Arm C: Investigator's Choice
Number analyzed (Participants) | 83 | 86 | 85
score on a scale
  Body Image (Week 1 Day 1): number analyzed (Participants) | 74 | 80 | 69
  Body Image (Week 1 Day 1) | 76.2 [0 to 100] | 80.1 [0 to 100] | 75.8 [0 to 100]
  Body Image (Week 7 Day 1): number analyzed (Participants) | 52 | 47 | 36
  Body Image (Week 7 Day 1) | 76.4 [11 to 100] | 77.6 [33 to 100] | 78.2 [0 to 100]
  Anxiety (Week 1 Day 1): number analyzed (Participants) | 74 | 81 | 69
  Anxiety (Week 1 Day 1) | 50.0 [0 to 100] | 48.2 [0 to 100] | 43.0 [0 to 100]
  Anxiety (Week 7 Day 1): number analyzed (Participants) | 52 | 48 | 36
  Anxiety (Week 7 Day 1) | 57.1 [0 to 100] | 61.1 [0 to 100] | 50.9 [0 to 100]
  Weight (Week 1 Day 1): number analyzed (Participants) | 73 | 81 | 69
  Weight (Week 1 Day 1) | 79.5 [0 to 100] | 85.6 [0 to 100] | 78.3 [0 to 100]
  Weight (Week 7 Day 1): number analyzed (Participants) | 52 | 48 | 36
  Weight (Week 7 Day 1) | 86.6 [33 to 100] | 89.6 [33 to 100] | 88.0 [0 to 100]
  Sexual Function (Men) (Week 1 Day 1): number analyzed (Participants) | 45 | 47 | 41
  Sexual Function (Men) (Week 1 Day 1) | 31.7 [0 to 100] | 21.2 [0 to 100] | 23.5 [0 to 100]
  Sexual Function (Men) (Week 7 Day 1): number analyzed (Participants) | 30 | 25 | 21
  Sexual Function (Men) (Week 7 Day 1) | 33.2 [0 to 100] | 26.6 [0 to 67] | 34.9 [0 to 100]
  Sexual Function (Women) (Week 1 Day 1): number analyzed (Participants) | 24 | 27 | 23
  Sexual Function (Women) (Week 1 Day 1) | 16.5 [0 to 33] | 12.3 [0 to 67] | 10.1 [0 to 67]
  Sexual Function (Women) (Week 7 Day 1): number analyzed (Participants) | 16 | 17 | 15
  Sexual Function (Women) (Week 7 Day 1) | 16.6 [0 to 67] | 13.6 [0 to 67] | 11.0 [0 to 33]
  Urinary Frequency (Week 1 Day 1): number analyzed (Participants) | 75 | 80 | 68
  Urinary Frequency (Week 1 Day 1) | 34.4 [0 to 100] | 30.3 [0 to 83] | 32.6 [0 to 100]
  Urinary Frequency (Week 7 Day 1): number analyzed (Participants) | 52 | 48 | 35
  Urinary Frequency (Week 7 Day 1) | 28.2 [0 to 100] | 28.8 [0 to 67] | 18.5 [0 to 67]
  Blood and Mucus (Week 1 Day 1): number analyzed (Participants) | 74 | 81 | 67
  Blood and Mucus (Week 1 Day 1) | 4.1 [0 to 50] | 1.5 [0 to 33] | 2.0 [0 to 33]
  Blood and Mucus (Week 7 Day 1): number analyzed (Participants) | 52 | 49 | 36
  Blood and Mucus (Week 7 Day 1) | 2.6 [0 to 33] | 3.1 [0 to 67] | 2.3 [0 to 33]
  Stool Frequency (Week 1 Day 1): number analyzed (Participants) | 55 | 68 | 57
  Stool Frequency (Week 1 Day 1) | 15.5 [0 to 100] | 11.3 [0 to 100] | 14.1 [0 to 83]
  Stool Frequency (Week 7 Day 1): number analyzed (Participants) | 40 | 41 | 32
  Stool Frequency (Week 7 Day 1) | 13.4 [0 to 50] | 11.8 [0 to 83] | 13.1 [0 to 67]
  Urinary Incontinence (Week 1 Day 1): number analyzed (Participants) | 73 | 79 | 67
  Urinary Incontinence (Week 1 Day 1) | 8.2 [0 to 100] | 7.5 [0 to 100] | 7.4 [0 to 100]
  Urinary Incontinence (Week 7 Day 1): number analyzed (Participants) | 52 | 48 | 35
  Urinary Incontinence (Week 7 Day 1) | 7.0 [0 to 67] | 4.8 [0 to 67] | 1.9 [0 to 33]
  Dysuria (Week 1 Day 1): number analyzed (Participants) | 75 | 80 | 66
  Dysuria (Week 1 Day 1) | 4.0 [0 to 33] | 2.9 [0 to 67] | 3.0 [0 to 67]
  Dysuria (Week 7 Day 1): number analyzed (Participants) | 51 | 48 | 35
  Dysuria (Week 7 Day 1) | 3.2 [0 to 33] | 2.1 [0 to 33] | 0.9 [0 to 33]
  Abdominal Pain (Week 1 Day 1): number analyzed (Participants) | 74 | 80 | 68
  Abdominal Pain (Week 1 Day 1) | 18.8 [0 to 100] | 12.8 [0 to 100] | 23.0 [0 to 100]
  Abdominal Pain (Week 7 Day 1): number analyzed (Participants) | 51 | 49 | 36
  Abdominal Pain (Week 7 Day 1) | 10.4 [0 to 67] | 10.8 [0 to 67] | 16.6 [0 to 67]
  Buttock Pain (Week 1 Day 1): number analyzed (Participants) | 74 | 80 | 67
  Buttock Pain (Week 1 Day 1) | 11.6 [0 to 100] | 10.8 [0 to 100] | 9.9 [0 to 100]
  Buttock Pain (Week 7 Day 1): number analyzed (Participants) | 52 | 49 | 36
  Buttock Pain (Week 7 Day 1) | 4.4 [0 to 33] | 8.8 [0 to 67] | 7.4 [0 to 67]
  Bloated Feeling (Week 1 Day 1): number analyzed (Participants) | 73 | 81 | 69
  Bloated Feeling (Week 1 Day 1) | 20.4 [0 to 100] | 14.8 [0 to 67] | 21.7 [0 to 100]
  Bloated Feeling (Week 7 Day 1): number analyzed (Participants) | 52 | 49 | 36
  Bloated Feeling (Week 7 Day 1) | 13.3 [0 to 67] | 12.1 [0 to 33] | 12.9 [0 to 67]
  Dry Mouth (Weel 1 Day 1): number analyzed (Participants) | 74 | 80 | 69
  Dry Mouth (Weel 1 Day 1) | 25.1 [0 to 100] | 17.0 [0 to 67] | 22.1 [0 to 100]
  Dry Mouth (Weel 7 Day 1): number analyzed (Participants) | 52 | 49 | 36
  Dry Mouth (Weel 7 Day 1) | 26.8 [0 to 100] | 29.2 [0 to 100] | 13.8 [0 to 67]
  Hair Loss (Week 1 Day 1): number analyzed (Participants) | 72 | 81 | 66
  Hair Loss (Week 1 Day 1) | 17.1 [0 to 100] | 11.1 [0 to 100] | 14.6 [0 to 100]
  Hair Loss (Week 7 Day 1): number analyzed (Participants) | 52 | 48 | 36
  Hair Loss (Week 7 Day 1) | 7.0 [0 to 100] | 7.6 [0 to 67] | 4.6 [0 to 100]
  Trouble with Taste (Week 1 Day 1): number analyzed (Participants) | 73 | 81 | 66
  Trouble with Taste (Week 1 Day 1) | 20.0 [0 to 100] | 13.9 [0 to 100] | 15.1 [0 to 100]
  Trouble with Taste (Week 7 Day 1): number analyzed (Participants) | 52 | 48 | 36
  Trouble with Taste (Week 7 Day 1) | 18.5 [0 to 100] | 15.2 [0 to 67] | 12.9 [0 to 100]
  Flatulence (Week 1 Day 1): number analyzed (Participants) | 56 | 68 | 56
  Flatulence (Week 1 Day 1) | 18.3 [0 to 100] | 19.5 [0 to 100] | 23.1 [0 to 100]
  Flatulence (Week 7 Day 1): number analyzed (Participants) | 40 | 41 | 32
  Flatulence (Week 7 Day 1) | 12.4 [0 to 67] | 16.1 [0 to 67] | 12.4 [0 to 33]
  Faecal Incontinence (Week 1 Day 1): number analyzed (Participants) | 56 | 68 | 56
  Faecal Incontinence (Week 1 Day 1) | 8.9 [0 to 100] | 8.8 [0 to 100] | 7.1 [0 to 67]
  Faecal Incontinence (Week 7 Day 1): number analyzed (Participants) | 40 | 41 | 32
  Faecal Incontinence (Week 7 Day 1) | 2.5 [0 to 33] | 7.3 [0 to 67] | 3.1 [0 to 33]
  Sore Skin (Week 1 Day 1): number analyzed (Participants) | 55 | 68 | 55
  Sore Skin (Week 1 Day 1) | 9.6 [0 to 67] | 8.8 [0 to 67] | 6.0 [0 to 33]
  Sore Skin (Week 7 Day 1): number analyzed (Participants) | 40 | 41 | 32
  Sore Skin (Week 7 Day 1) | 11.6 [0 to 33] | 9.7 [0 to 67] | 4.2 [0 to 67]
  Embarrassed by Bowel Movement (Week 1 Day 1): number analyzed (Participants) | 55 | 68 | 55
  Embarrassed by Bowel Movement (Week 1 Day 1) | 8.5 [0 to 100] | 7.8 [0 to 100] | 13.9 [0 to 100]
  Embarrassed by Bowel Movement (Week 7 Day 1): number analyzed (Participants) | 40 | 41 | 32
  Embarrassed by Bowel Movement (Week 7 Day 1) | 7.5 [0 to 67] | 8.1 [0 to 67] | 10.4 [0 to 67]
  Stoma Care Problem (Week 1 Day 1): number analyzed (Participants) | 16 | 20 | 25
  Stoma Care Problem (Week 1 Day 1) | 16.6 [0 to 100] | 3.3 [0 to 33] | 6.6 [0 to 67]
  Stoma Care Problem (Week 7 Day 1): number analyzed (Participants) | 10 | 14 | 8
  Stoma Care Problem (Week 7 Day 1) | 9.9 [0 to 33] | 2.4 [0 to 33] | 8.3 [0 to 33]
  Impotence (Week 1 Day 1): number analyzed (Participants) | 44 | 43 | 41
  Impotence (Week 1 Day 1) | 46.9 [0 to 100] | 38.7 [0 to 100] | 49.5 [0 to 100]
  Impotence (Week 7 Day 1): number analyzed (Participants) | 28 | 25 | 21
  Impotence (Week 7 Day 1) | 40.4 [0 to 100] | 42.7 [0 to 100] | 50.7 [0 to 100]
  Dyspareunia (Week 1 Day 1): number analyzed (Participants) | 22 | 23 | 21
  Dyspareunia (Week 1 Day 1) | 12.1 [0 to 100] | 7.2 [0 to 33] | 11.0 [0 to 100]
  Dyspareunia (Week 7 Day 1): number analyzed (Participants) | 14 | 16 | 15
  Dyspareunia (Week 7 Day 1) | 14.3 [0 to 67] | 10.3 [0 to 33] | 13.3 [0 to 67]

12. Secondary Outcome: Quality of Life Assessed by FACT-EGFRI-18 for Skin Rash
Description: Scale: Functional Assessment of Cancer Therapy-Epidermal Growth Factor Receptor Inhibitor 18 (FACT-EGFRI-18).
  The FACT-EGFRI-18 is an 18-question scale used to assess EGFR-inhibitor-treated cancer patients' quality of life relative to their experience of skin rash based on three (3) multi-item subscales. The subscales combined (i.e., Symptom Index) range in score from 0 to 72. A higher score represents a high level of symptomatology (problems).
  High scores for all subscales represent a worse outcome:
  * The Physical subscale ranges in score from 0 to 28.
  * The Social/Emotional subscale ranges in score from 0 to 24.
  * The Functional subscale ranges in score from 0 to 20.
Time Frame: Assessed every 3 weeks (week 1 and week 4 reported)
Population: This measure was self-reported. Numbers analyzed between Week 1 and Week 4 differ from each other, as well from the overall number of subjects analyzed. Data could not be collected from subjects not compliant with reporting or once discontinued.
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Arm A: Sym004 (12 mg/kg) | Arm B: Sym004 (9/6 mg/kg) | Arm C: Investigator's Choice
Number analyzed (Participants) | 83 | 86 | 85
score on a scale
  Physical (Week 1 Day 1): number analyzed (Participants) | 70 | 78 | 68
  Physical (Week 1 Day 1) | 22.9 [2 to 28] | 23.1 [4 to 28] | 24.3 [6 to 28]
  Physical (Week 4 Day 1): number analyzed (Participants) | 68 | 70 | 58
  Physical (Week 4 Day 1) | 18.0 [4 to 28] | 19.7 [5 to 28] | 25.1 [16 to 28]
  Social/Emotional (Week 1 Day 1): number analyzed (Participants) | 70 | 78 | 68
  Social/Emotional (Week 1 Day 1) | 21.5 [9 to 24] | 21.5 [6 to 24] | 22.6 [9 to 24]
  Social/Emotional (Week 4 Day 1): number analyzed (Participants) | 68 | 70 | 58
  Social/Emotional (Week 4 Day 1) | 19.9 [7 to 24] | 20.3 [5 to 24] | 23.2 [15 to 24]
  Functional (Week 1 Day 1): number analyzed (Participants) | 70 | 78 | 68
  Functional (Week 1 Day 1) | 17.9 [5 to 20] | 18.3 [7 to 20] | 18.7 [4 to 20]
  Functional (Week 4 Day 1): number analyzed (Participants) | 68 | 70 | 58
  Functional (Week 4 Day 1) | 16.3 [3 to 20] | 17.0 [6 to 20] | 19.3 [13 to 20]
  Symptom Index (Week 1 Day 1): number analyzed (Participants) | 70 | 78 | 68
  Symptom Index (Week 1 Day 1) | 62.3 [18 to 72] | 62.9 [20 to 72] | 65.6 [19 to 72]
  Symptom Index (Week 4 Day 1): number analyzed (Participants) | 68 | 70 | 58
  Symptom Index (Week 4 Day 1) | 54.2 [16 to 72] | 57.0 [22 to 72] | 67.6 [46 to 72]

13. Post Hoc Outcome: Overall Survival (OS) Time for Patients in Europe + United States With Double-Negative mCRC (EU+US DNmCRC)
Description: OS based on product-limit (Kaplan-Meier) estimates. Confidence intervals for the median are calculated according to Brookmeyer and Crowley.
  This outcome measure is considered exploratory. Because of the unanticipated long OS in the control group, initial exploratory subgroup analyses identified that findings in patients enrolled in Russia differed when compared with patients enrolled in the ITT subpopulation and the EU+US subpopulation. For this reason, subjects in Russia were excluded from further exploratory subset analyses that evaluated the effects of genomic parameters known to impact patient responses to anti-EGFR monoclonal antibodies. Removal of the outlier Russian subpopulation of patients provided a patient population that was more homogeneous with respect to their prior treatment regimens, thereby facilitating further exploratory analyses. If a subject had not died, survival time was censored at the last date the subject was known to be alive.
Time Frame: From randomization until the date of death (assessed up to 32 months).
Population: The analysis population was the EU+US DNmCRC analysis set, which is a genomically-defined subpopulation excluding patients with high frequency clonal RAS mutations and BRAF V600E mutations.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A: Sym004 (12 mg/kg) | Arm B: Sym004 (9/6 mg/kg) | Arm C: Investigator's Choice
Number analyzed (Participants) | 62 | 57 | 51
months | 8.9 [6.2 to 12.4] | 11.9 [9.7 to 13.8] | 8.4 [6.4 to 10.0]

14. Post Hoc Outcome: Overall Survival (OS) Time for Patients in Europe + United States With Triple-Negative mCRC (EU+US TNmCRC)
Description: as for outcome 13
Time Frame: From randomization until the date of death (assessed up to 32 months).
Population: The analysis population was the EU+US TNmCRC analysis set, which is a genomically-defined subpopulation excluding DNmCRC patients with six (6) selected EGFR extracellular domain (ECD) mutations.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A: Sym004 (12 mg/kg) | Arm B: Sym004 (9/6 mg/kg) | Arm C: Investigator's Choice
Number analyzed (Participants) | 47 | 46 | 38
months | 10.6 [6.8 to 13.1] | 12.8 [9.7 to 14.7] | 7.3 [6.3 to 8.8]

ADVERSE EVENTS:
Time Frame: Adverse event (AE) data were collected beginning with the signing of informed consent and continued through the End of Trial Intervention Visit (i.e., no earlier than 28 days after stop of treatment). The AE data collection period was 38 months.
Description: Subjects analyzed for the Serious Adverse Events and Other (Not Including Serious) Adverse Events tables are based on the Safety Analysis Set. The Safety Analysis Set contained all subjects in the Intent-to-Treat (ITT) Analysis Set who received at least one (1) dose of trial treatment (Sym004, 5-FU, or capecitabine) and in addition, those subjects who received Best Supportive Care only. The All-Cause Mortality table also includes those subjects who were randomized but not treated.
Arm/Group | Arm A: Sym004 (12 mg/kg) | Arm B: Sym004 (9/6 mg/kg) | Arm C: Investigator's Choice
All-Cause Mortality (participants affected / at risk) | 68/83 | 62/86 | 57/85
Serious Adverse Events (participants affected / at risk) | 27/83 | 23/84 | 12/78
Other Adverse Events (participants affected / at risk) | 83/83 | 84/84 | 67/78
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A: Sym004 (12 mg/kg) (N=83) | Arm B: Sym004 (9/6 mg/kg) (N=84) | Arm C: Investigator's Choice (N=78)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Acute coronary syndrome (Cardiac disorders) | 0 | 1 | 0
Cardiac arrest (Cardiac disorders) | 0 | 0 | 1
Cardiac failure (Cardiac disorders) | 0 | 0 | 1
Sinus node dysfunction (Cardiac disorders) | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 1 | 2
Intestinal obstruction (Gastrointestinal disorders) | 2 | 2 | 1
Vomiting (Gastrointestinal disorders) | 2 | 0 | 3
Colitis (Gastrointestinal disorders) | 0 | 0 | 1
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0 | 0
Rectal obstruction (Gastrointestinal disorders) | 1 | 0 | 0
Pyrexia (General disorders) | 2 | 2 | 0
Asthenia (General disorders) | 1 | 1 | 0
General physical health deterioration (General disorders) | 2 | 0 | 0
Oedema peripheral (General disorders) | 0 | 2 | 0
Chest pain (General disorders) | 0 | 1 | 0
Hyperthermia (General disorders) | 1 | 0 | 0
Jaundice cholestatic (Hepatobiliary disorders) | 0 | 1 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 0 | 0
Hepatorenal syndrome (Hepatobiliary disorders) | 1 | 0 | 0
Device related infection (Infections and infestations) | 1 | 2 | 1
Pneumonia (Infections and infestations) | 2 | 1 | 0
Sepsis (Infections and infestations) | 1 | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 1 | 0
Abdominal abscess (Infections and infestations) | 0 | 0 | 1
Bacteraemia (Infections and infestations) | 0 | 0 | 1
Device related sepsis (Infections and infestations) | 0 | 1 | 0
Impetigo (Infections and infestations) | 1 | 0 | 0
Staphylococcal sepsis (Infections and infestations) | 0 | 0 | 1
Urosepsis (Infections and infestations) | 1 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 2 | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Urinary tract stoma complication (Injury, poisoning and procedural complications) | 1 | 0 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 4 | 5 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Seizure (Nervous system disorders) | 1 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 1 | 1
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 1
Renal failure (Renal and urinary disorders) | 0 | 1 | 0
Vesicocutaneous fistula (Renal and urinary disorders) | 0 | 0 | 1
Pelvic pain (Reproductive system and breast disorders) | 0 | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Blister (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Skin toxicity (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A: Sym004 (12 mg/kg) (N=83) | Arm B: Sym004 (9/6 mg/kg) (N=84) | Arm C: Investigator's Choice (N=78)
Anaemia (Blood and lymphatic system disorders) | 10 | 15 | 11
Thrombocytopenia (Blood and lymphatic system disorders) | 3 | 7 | 8
Leukopenia (Blood and lymphatic system disorders) | 4 | 7 | 5
Neutropenia (Blood and lymphatic system disorders) | 2 | 4 | 9
Sinus tachycardia (Cardiac disorders) | 7 | 11 | 7
Supraventricular extrasystoles (Cardiac disorders) | 1 | 5 | 2
Diarrhoea (Gastrointestinal disorders) | 10 | 19 | 20
Abdominal pain (Gastrointestinal disorders) | 13 | 10 | 3
Nausea (Gastrointestinal disorders) | 9 | 10 | 12
Vomiting (Gastrointestinal disorders) | 6 | 4 | 6
Constipation (Gastrointestinal disorders) | 6 | 3 | 6
Stomatitis (Gastrointestinal disorders) | 8 | 4 | 0
Abdominal pain upper (Gastrointestinal disorders) | 2 | 0 | 4
Asthenia (General disorders) | 26 | 21 | 14
Xerosis (General disorders) | 26 | 12 | 0
Pyrexia (General disorders) | 12 | 10 | 9
Fatigue (General disorders) | 8 | 7 | 14
Oedema peripheral (General disorders) | 9 | 7 | 1
Mucosal inflammation (General disorders) | 8 | 6 | 4
Chills (General disorders) | 3 | 5 | 1
Paronychia (Infections and infestations) | 15 | 18 | 3
Conjunctivitis (Infections and infestations) | 13 | 8 | 1
Urinary tract infection (Infections and infestations) | 5 | 3 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 5 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 18 | 15 | 0
Blood alkaline phosphatase increased (Investigations) | 7 | 10 | 6
Alanine aminotransferase increased (Investigations) | 7 | 8 | 0
Aspartate aminotransferase increased (Investigations) | 8 | 6 | 1
Electrocardiogram QT prolonged (Investigations) | 6 | 7 | 2
Blood bilirubin increased (Investigations) | 5 | 2 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 57 | 47 | 6
Decreased appetite (Metabolism and nutrition disorders) | 20 | 9 | 7
Hypocalcaemia (Metabolism and nutrition disorders) | 9 | 8 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 10 | 4 | 3
Hyperglycaemia (Metabolism and nutrition disorders) | 4 | 5 | 2
Hypoalbuminaemia (Metabolism and nutrition disorders) | 3 | 5 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 5 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 5 | 5 | 7
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3 | 5 | 1
Insomnia (Psychiatric disorders) | 9 | 2 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 | 3 | 6
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 5 | 5
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 68 | 65 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 33 | 30 | 2
Skin fissures (Skin and subcutaneous tissue disorders) | 14 | 16 | 2
Erythema (Skin and subcutaneous tissue disorders) | 16 | 11 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 8 | 10 | 1
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 | 1 | 14
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 10 | 4 | 0
Rash (Skin and subcutaneous tissue disorders) | 7 | 6 | 0
Hypertension (Vascular disorders) | 6 | 2 | 1

LIMITATIONS AND CAVEATS:
Considering the hypothesis-generating nature of a phase 2 clinical trial, the intent-to-treat (ITT) analysis should be viewed as the starting point of a scientific investigation process, not the final conclusion.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator will inform the sponsor in advance about any plans to publish or present data from the trial. Any publications and presentations of the results (abstracts in journals or newspapers, oral presentations, etc.), either in whole or in part, by investigators or their representatives will require pre-submission review by the sponsor. The sponsor will not suppress or veto publications, but maintains the right to delay publication in order to protect intellectual property rights.